CLINICAL TRIAL: NCT00002586
Title: ASSESSMENT OF INTERMEDIATE ENDPOINT BIOMARKERS TO 13-CIS RETINOIC ACID WITH OR WITHOUT ALPHA TOCOPHEROL OR OBSERVATION
Brief Title: 13-Cis Retinoic Acid With or Without Vitamin E for Prevention of Lung Cancer
Acronym: 13-Cis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 92-0382; NCI-V94-0506 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Drug Toxicity; Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Isotretinoin; Tocopherols; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 13-cis retinoic acid (Experimental): 13-cis retinoic acid 50 mg/d
  Interventions: Drug: 13-cis retinoic acid
- 13-Cis Retinoic Acid and Tocopherol (Experimental): 13-Cis Retinoic Acid (50 mg/day) Tocopherol (800 mg/day)
  Interventions: Drug: 13-cis retinoic acid; Dietary Supplement: Tocopherol
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: 13-cis retinoic acid
  Other Names: Isotretinoin, AccutaneT
  Arms: 13-Cis Retinoic Acid and Tocopherol; 13-cis retinoic acid
Dietary Supplement: Tocopherol
  Other Names: Vitamin E
  Arms: 13-Cis Retinoic Acid and Tocopherol

SUMMARY:
RATIONALE: 13 Cis retinoic acid may prevent the development of cancer cells.

PURPOSE: Randomized double-blinded phase II trial to study the effectiveness of 13-cis retinoic acid with or without vitamin E for chemoprevention or observation of cancer in persons at high risk of developing lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if alpha tocopherol can reduce the toxicities of low dose 13-cis retinoic acid administered for one year.
* To access the adequacy of the collected specimens for studies of intermediate endpoint markers.
* to establish a depository of biologic specimens for future studies of new biomarkers.

  * Arm 1: Patients receive oral 13-cis retinoic acid daily.
  * Arm 2: Patients receive oral 13-cis retinoic acid and oral vitamin E daily.
  * Arm 3: Patients undergo observation only. Treatment continues in arms I and II for 1 year in the absence of unacceptable toxicity.

Patients are followed annually for 2 years.

PROJECTED ACCRUAL: A total of 100 patients (33 Arm 1, 33 Arm 2, and 34 Arm 3) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients identified through the Tissue Procurement/Screening Project with mild, moderate or severe dysplasia, Ca In situ OR surgically cured patients with head and neck cancer who are found to have mild atypia or greater on their staging bronchoscopy. (This includes carcinoma in situ). Also eligible are patients with Stage I and II non-small cell lung cancer who are disease free greater than 36 months.
2. Patients must have at least a 30 pack year smoking history.
3. Patients must be a current smoker or ex-smoker who have not smoked for at least 6 months more.
4. Patients must have peripheral granulocyte count of > 1500 and platelet count of > 150,000.
5. Patients must have adequate hepatic function with bilirubin < 1.5 mg % and SGPT < 4 times institutional upper limits of normal.
6. Patients must have adequate renal function with serum creatinine < 1.5 mg %.
7. All patients must be informed of the investigational nature of the study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Patients must not have a current or past history of cancer within the past 5 years with the exception of surgically cured head and neck cancer or surgically cured Stage I or II lung cancer > 36 months from diagnosis or skin cancer or in situ cancers.
2. Patients must have no serious intercurrent illness including insulin dependent diabetes mellitus or hypercholesterolemia (>239mg/dl) / hypertriglyceridemia (>149mg/dl).
3. Patients must not have evidence of clinically active coronary artery disease including myocardial infarction within 6 weeks, chest pain or poorly controlled congestive heart failure or any other serious medical condition, which would preclude a patient from undergoing a bronchoscopy.
4. Patients must not have cardiac dysrhythmia that is potentially life threatening such as ventricular tachycardia, multifocal premature ventricular contractions or supraventricular tachycardias with a rapid ventricular response. Well controlled atrial fibrillation or rare (<2/minute) premature ventricular contractions are not exclusionary
5. Chest x-ray must not show evidence of tumor.
6. Patients must not be taking vitamin A or E supplements
7. Patients must not be taking tetracycline or minocycline.
8. Patients who have had prior chemotherapy or radiation therapy.
9. Women who are pregnant are ineligible

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 1993-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Treatment failure | Three years
  Treatment "failure" defined as histologic progression (any increase in the maximum histologic score) or failure to return for follow-up bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: York E. Miller, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - National Jewish Center for Immunology and Respiratory Medicine, Denver, Colorado
  - Lung Cancer Institute, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado

REFERENCES:
- [Result] Kelly K, Kittelson J, Franklin WA, Kennedy TC, Klein CE, Keith RL, Dempsey EC, Lewis M, Jackson MK, Hirsch FR, Bunn PA, Miller YE. A randomized phase II chemoprevention trial of 13-CIS retinoic acid with or without alpha tocopherol or observation in subjects at high risk for lung cancer. Cancer Prev Res (Phila). 2009 May;2(5):440-9. doi: 10.1158/1940-6207.CAPR-08-0136. Epub 2009 Apr 28. PMID 19401528